CLINICAL TRIAL: NCT04688203
Title: Effects of Magnesium Sulfate and Labetalol Infusion Used for Induced Hypotension on Peripheral Perfusion and Postoperative Pain in Nasal Surgeries
Brief Title: Effects Magnesium Sulfate and Labetalol Infusion on Peripheral Perfusion and Pain in Nasal Surgeries
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Alshaimaa Abdel Fattah Kamel, lecturer of Anesthesia ,and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6601
Record Dates: First submitted 2020-12-20; First posted 2020-12-29 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Peripheral Perfusion; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium Sulfate; Labetalol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium sulfate infudsion (Active Comparator): patients will receive IV bolus dose of 40mg/kg magnesium sulfate in 100 ml saline solution over ten minutes then continuous infusion of 10-15mg/kg/h will be titrated till achieve target mean arterial blood pressure (55-65 mmHg) and will be terminated by the end of surgery.
  Interventions: Drug: Magnesium Sulfate Injection
- Labetalol infusion (Active Comparator): will receive IV bolus does of labetalol 0.25 mg/kg over ten minutes then continuous infusion of 0.5-1mg/kg/h will be titrated till achieve target mean arterial blood pressure (55-65 mmHg) and will be terminated by the end of surgery.
  Interventions: Drug: Labetalol Injectable Solution

INTERVENTIONS:
Drug: Magnesium Sulfate Injection — will receive IV bolus dose of 40mg/kg magnesium sulfate in 100 ml saline solution over ten minutes then continuous infusion of 10-15mg/kg/h will be titrated till achieve target mean arterial blood pressure (55-65 mmHg) and will be terminated by the end of surgery.
  Other Names: magnesium sulfate
  Arms: Magnesium sulfate infudsion
Drug: Labetalol Injectable Solution — will receive IV bolus does of labetalol 0.25 mg/kg over ten minutes then continuous infusion of 0.5-1mg/kg/h will be titrated till achieve target mean arterial blood pressure (55-65 mmHg) and will be terminated by the end of surgery.
  Other Names: labetalol
  Arms: Labetalol infusion

SUMMARY:
One of main risk of controlled hypotension during nasal surgeries is impaired perfusion. Peripheral perfusion of non-vital organs usually impaired earlier than vital organs. So, evaluation of perfusion of non-vital organ is considered to be adequate measure of patient safety during surgery.

Many hypotensive agents such as dexmedetomidine, B blockers, magnesium sulfate and nitroglycerine had been used but we are in need to investigate its effects on peripheral perfusion.

Postoperative pain related to nasal surgeries due to surgical trauma itself which induces the release of inflammatory mediators from neuronal and immune cells resulting in peripheral and central sensitization significantly affects recovery of patients. Magnesium sulfate and labetalol have analgesic actions besides their hypotensive effects but with different mechanisms.

DETAILED DESCRIPTION:
To compare between the effects of magnesium sulfate and labetalol infusion during induced hypotension on peripheral perfusion and postoperative pain in nasal surgeries

OBJECTIVES:

To measure peripheral perfusion index (PPI) as an indicator for peripheral perfusion To calculate the total postoperative rescue analgesic requirements.

Double -blind randomized comparative Clinical Study. All Patients will be randomly allocated into two equal groups (group M and Group L).

Using computer generated randomization table, each group will be 25 patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient.
* Age: 21-45 years old.
* Sex: both sex (males or females).
* Physical status: ASA 1& II.
* BMI = (20-30 kg/m2).
* Type of operations: elective nasal surgeries such as septoplasty, endoscopic sinus surgery and polypectomy.
* Duration of surgery ≤ two hours.

Exclusion Criteria:

* Altered mental state
* Patients on beta blocker or with known history of allergy to study drugs.
* Advanced hepatic, renal, cardiovascular or respiratory diseases.
* Diabetic patients.
* Patients receiving anticoagulants or on pain killers.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Peripheral perfusion index | Changes from baseline Peripheral perfusion index at 2 hours.
  Peripheral perfusion index by pulse oximertry will be measured at basal, 3minutes after induction, every 10 minutes till end of surgery. It will be calculated by dividing the pulsatile signal to nonpulsatile. The normal range is (0.02% -20%)

SECONDARY OUTCOMES:
Mean arterial blood pressure | basal then at 3 minutes after intubation, and after skin incision then every 10 minutes till the end of surgery
  Mean arterial blood pressure will be recorded at basal, 3 minutes after intubation, and after skin incision then every 10 min till the end of surgery.
Heart rate | basal then at 3 minutes after intubation, and after skin incision then every 10 minutes till the end of surgery
  Heart rate will be recorded at basal, 3 minutes after intubation, and after skin incision then every 10 min till the end of surgery.
postoperative Pain intensity | at 30 minutes, 1 hour, 2hours, 4hours, 6hours, 12hours, and 24hours postoperative.
  Postoperative Pain will be assessed using Numerical rating Scale (NRS) . A commonly used scale is a 10-cm line labeled with "worst pain imaginable" on the right border and "no pain" on the left border. The patient will be instructed to make a mark along the line to represent the intensity of pain currently being experienced. NRS score 4 or more =pain. Paracetamol 1gm IV will be given every 6 hours as a protocol for pain management will be started at the end of surgery, and IV pethidine 1mg/kg (rescue analgesic) will be given if NRS >4.
time to first call for pethidine (rescue analgesic) | up to 24hour postoperative
  Time from the stoppage of infusion solution to first call for pethidine (rescue analgesic) will be recorded.
Total pethidine requirements | up to 24hour postoperative
  Total pethidine requirements
Serum lactate level | basal and at one hour after extubation
  Serum lactate will be recorded basal and at one hour after extubation. The normal serum lactate ranges from 4.5 to 19.8 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa Kamel, M.D, Principal Investigator — Faculty of Human medicine, Zagazig university
Locations (1):
- Alshaimaa Abdel Fattah Kamel, Zagazig, Egypt

REFERENCES:
- [Derived] Kamel AAF, Medhat MM, Salem DAE, Naby SMA. Effect of perioperative magnesium sulfate and labetalol infusion on peripheral perfusion and postoperative pain in nasal surgery: a randomized controlled trial. Patient Saf Surg. 2022 Aug 19;16(1):27. doi: 10.1186/s13037-022-00336-7. PMID 35986325